CLINICAL TRIAL: NCT06212427
Title: Feeding Tolerance and Growth of Preterm Infants Consuming a Supplement Containing Two Human Milk Oligosaccharides (HMOs): A Post-Market Study
Brief Title: Feeding Tolerance and Growth of Preterm Infants Consuming a Supplement Containing Two Human Milk Oligosaccharides (HMOs)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2211INF
Record Dates: First submitted 2023-12-07; First posted 2024-01-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Premature Infant; Low Birthweight Infant
Keywords: Human Milk Oligosaccharides; Feeding tolerance; Growth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMO supplement (Other)
  Interventions: Dietary Supplement: HMO supplement

INTERVENTIONS:
Dietary Supplement: HMO supplement — Liquid supplement containing 2 specific HMOs. Supplement will be given 3-4 times a day, not mixed with any feeding.

SUMMARY:
The goal of this post-market study is to describe the effect of a liquid supplement containing 2 specific human milk oligosaccharides (HMOs), 2'-fucosyllactose [2'FL] and lacto-N-neotetraose [LNnT], on feeding tolerance, growth, and adverse events of special interest in preterm infants in a real-world setting.

A comparison with data collected retrospectively from a historical group at each site will be made for time to reach full enteral feeding, growth and adverse events. Infants in the historical group were not exposed to an HMO supplement but followed the same local nutrition protocol to avoid confounding by differences in clinical or feeding practice.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from at least one parent (or other legally acceptable representative [LAR], if applicable)
2. Infant's parent(s)/LAR is of legal age of majority, has parental authority, must understand the consent form and other relevant study documents, and is willing and able to fulfil the requirements of the study protocol
3. Infant gestational age is ≤ 34 weeks as determined by the first day of the mother's last menstrual period or by fetal ultrasound
4. Infant birth weight ≤ 2500g
5. Infant postnatal age ≤ 14 days
6. Infant has tolerated trophic feeds (e.g., 10-15 mL/kg/day) for at least 24 hours but has not yet reached full enteral feeding

Exclusion Criteria:

1. Infant is clinically unstable, for example:

   1. Infant has hemodynamic instability as evidenced by clinical signs of sepsis, hypotension (MAP < 5th percentile for age for at least three hours), or is receiving vasopressor drugs
   2. Infant has received an exchange transfusion within the past 48 hours
   3. Infant has had an episode of severe asphyxia at birth (PH less than 7.0)
   4. Infant has signs of necrotizing enterocolitis according to modified Bell staging criteria (stage IIA or higher)
2. Major congenital (e.g., heart disease, skeletal dysplasia, chondrodystrophy, gastrointestinal obstruction or atresia) or chromosomal abnormality (e.g., trisomy 21, Turner syndrome)
3. Infant has other medical condition that, in the judgement of the investigator, would make the child inappropriate for entry into the study
4. Participation in another interventional clinical study that may interfere with the results of this study

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Feeding tolerance | From birth until achievement of full enteral feeding (1 to 3 weeks)
  Time to reach full enteral feeding rate of 150 mL/kg/day
Feeding tolerance | From birth until achievement of full enteral feeding (1 to 3 weeks)
  Time to reach cessation of parenteral feeding

SECONDARY OUTCOMES:
Gastrointestinal tolerance | From enrollment (baseline) until NICU discharge (V5), assessed up to 13 weeks
  Through data collected from neonatal unit records
Weight gain | From enrollment (baseline) until NICU discharge (V5), assessed up to 13 weeks
  Measured in kilograms per day
Length gain | From enrollment (baseline) until NICU discharge (V5), assessed up to 13 weeks
  Measured in centimeters per week
Head circumference gain | From enrollment (baseline) until NICU discharge (V5), assessed up to 13 weeks
  Measured in centimeters per week
Safety via reporting of adverse events (AEs) and serious adverse events (SAEs) | From enrollment (baseline) until NICU discharge (V5), assessed up to 13 weeks
  Type, incidence, severity, seriousness, and relation to HMO supplement consumption as well as concomitant medications and non-pharmacological treatments.
  The incidence of specific illnesses of interest
  a. Necrotizing enterocolitis b Confirmed or suspected late-onset sepsis c. Bronchopulmonary dysplasia d. Retinopathy of prematurity

CONTACTS AND LOCATIONS:
Locations (6):
- Kepler Universitätsklinikum Linz, Linz, Austria
- Germany (5):
  - Evangelisches Waldkrankenhaus Spandau, Berlin-Spandau
  - Kinderklinik Darmstadt, Darmstadt
  - Wilhelmstift Hamburg, Hamburg
  - Uniklinik Heidelberg, Heidelberg
  - Klinikum Nürnberg, Nuremberg